CLINICAL TRIAL: NCT02628132
Title: Study of the Safety, Tolerability and Efficacy of the Investigational Anti PD-L1 Monoclonal Antibody Durvalumab in Combination With Paclitaxel in Patients With Metastatic Triple Negative PD-L1 Positive Breast Cancer
Brief Title: Study of Safety and Efficacy of Durvalumab in Combination With Paclitaxel in Metastatic Triple Negative Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2151-169; ESR-14-10649 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2015-11-29; First posted 2015-12-11 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: triple negative; breast cancer; durvalumab; paclitaxel; safety; efficacy; PD-L1; PD-1; Metastatic; AstraZeneca; MEDI4736
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Durvalumab and Paclitaxel (Experimental): After one cycle of paclitaxel, durvalumab will be given concurrently with paclitaxel. Once paclitaxel cycles are completed, durvalumab will be continued alone until disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Durvalumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel will be given weekly for 6 cycles
Drug: Durvalumab — Durvalumab will be given q2 wks concurrently with paclitaxel.
  Other Names: MEDI4736

SUMMARY:
The expression of PD-L1 in breast cancer has been previously demonstrated (Ghebeh et al 2006). In addition, PD-L1 has been shown to work as a "molecular shield", by protecting cancer cells from cytotoxic T-cells and chemotherapy induced apoptosis (Ghebeh et al 2008) suggesting to combine PD-L1 blockade with chemotherapy.

This trial will test Durvalumab in combination with Paclitaxel on metastatic triple-negative breast cancer patients. The safety profile of Durvalumab as a monotherapy has been previously established (lu et al 2015). In this trial the safety profile and tolerability of Durvalumab given in combination of Paclitaxel will be tested. In addition, the efficacy of this combination on metastatic breast cancer will be monitored.

DETAILED DESCRIPTION:
This open label single arm trial will involve metastatic triple negative PD-L1 positive breast cancer patients. The trial will include a dose deescalation phase where three doses of paclitaxel will be tried on 3 patients each followed by a dose expansion phase on 25 patients. Paclitaxel will be given weekly for 1 cycle followed by combination of Paclitaxel and Durvalumab. Once 6 cycles of Paclitaxel are completed, Durvalumab will be given alone until disease progression or unacceptable toxicity. The toxicity and tolerability of the combination will be the main end point while the efficacy will be a secondary end point.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed metastatic breast cancer
2. Triple negative breast cancer (estrogen receptor (ER) negative, progesterone receptor (PR) negative and Her2/neu negative).
3. Patients had received at least 1 line of chemotherapy in metastatic setting before being enrolled in this trial.
4. Written informed consent and any locally-required authorization
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Life expectancy of >12 weeks
7. Adequate normal organ and marrow functions.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study or previous enrolment in the present study
2. Participation in another clinical study with an investigational product during the last 4 months
3. Any previous treatment with a PD-1 or PD-L1 inhibitor, including MEDI4736 or with a CTLA 4 inhibitor
4. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
5. Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exceptions of 10 mg dexamethasone prior to paclitaxel infusion and intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
6. Active or prior documented autoimmune disease within the past 2 years
7. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
8. History of primary immunodeficiency
9. History of allogeneic organ transplant
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, interstitial lung disease (ILD), cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
11. Known history of previous clinical diagnosis of tuberculosis
12. History of leptomeningeal carcinomatosis
13. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving MEDI4736
14. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
15. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
16. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
17. Subjects with uncontrolled seizures.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events (severe and non-severe) | 12 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
Progression free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Ghebeh, B.Pharm, Ph.D., Principal Investigator — Research Center, King Faisal Specialist Hospital & Research Center; Taher Al-Tweigeri, M.D., Principal Investigator — Oncology Center, King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Ghebeh H, Mohammed S, Al-Omair A, Qattan A, Lehe C, Al-Qudaihi G, Elkum N, Alshabanah M, Bin Amer S, Tulbah A, Ajarim D, Al-Tweigeri T, Dermime S. The B7-H1 (PD-L1) T lymphocyte-inhibitory molecule is expressed in breast cancer patients with infiltrating ductal carcinoma: correlation with important high-risk prognostic factors. Neoplasia. 2006 Mar;8(3):190-8. doi: 10.1593/neo.05733. PMID 16611412
- [Background] Alsuliman A, Colak D, Al-Harazi O, Fitwi H, Tulbah A, Al-Tweigeri T, Al-Alwan M, Ghebeh H. Bidirectional crosstalk between PD-L1 expression and epithelial to mesenchymal transition: significance in claudin-low breast cancer cells. Mol Cancer. 2015 Aug 7;14:149. doi: 10.1186/s12943-015-0421-2. PMID 26245467
- [Background] Lu J, Lee-Gabel L, Nadeau MC, Ferencz TM, Soefje SA. Clinical evaluation of compounds targeting PD-1/PD-L1 pathway for cancer immunotherapy. J Oncol Pharm Pract. 2015 Dec;21(6):451-67. doi: 10.1177/1078155214538087. Epub 2014 Jun 9. PMID 24917416
- [Derived] Ghebeh H, Al-Sayed A, Eiada R, Cabangon L, Ajarim D, Suleman K, Tulbah A, Al-Tweigeri T. Weekly Paclitaxel given concurrently with Durvalumab has a favorable safety profile in triple-negative metastatic breast cancer. Sci Rep. 2021 Sep 27;11(1):19154. doi: 10.1038/s41598-021-98113-6. PMID 34580336